CLINICAL TRIAL: NCT06279676
Title: Improvement of Women's Health After Allogeneic Stem Cell Transplantation
Acronym: SaFeGreff
Status: Not yet recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: SaFeGreff
Record Dates: First submitted 2023-12-15; First posted 2024-02-28 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: GVHD, Chronic
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Human papilloma virus (HPV) sampling will be performed to assess reactivation and sub-types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective research project is to better understand vulvovaginal cGVHD to improve care of allografted women. The expected outcomes include better knowledge of the incidence and manifestations of vulvovaginal cGVHD, risk factors, response to treatments and impact on sexual health of allotransplanted female patients. The knowledge acquired will allow transplant clinicians to make more precise recommendations for gynecological management of future allografted women.

DETAILED DESCRIPTION:
The invetigators plan to recruit 100 women who will be evaluated 9 times over a period of 2 years (before allograft, at + 3 months, +6 months, +9 months, +12 months, +15 months, +18 months, +21 months, and +24 months +/- 14 days). If a new diagnosis of cGVHD is made between 2 visits, an additional gynecological examination will be performed.

Visits by the Hôpital Maisonneuve-Rosemont Hospital transplant team will include a physical examination to assess for the presence of cGVHD using the NIH criteria. The FACT-BMT quality of life questionnaire will also be completed before the allograft, at 3 months and 6 months after transplant. If cGVHD is diagnosed, the participants will also have to complete two questionnaires specific to cGVHD (Lee Scale for cGVHD, Patient self-assessment of cGVHD) at diagnosis and then at + 6, +12, +18 and +24 months from day 0 of allograft.

Assessments by CHUM gynecologists will take place before the allograft, then at +3, +6, +12, +18 and +24 months from day 0 of the allograft and will include: a vulvar/vaginal examination, a sample for HPV testing and sexual health questionnaires to be completed (Personal assessment of intimacy within relationships - PAIR, Female Sexual Function Index - FSFI , Female Sexual Distress Scale-Revised - FSDS-R).

ELIGIBILITY:
Inclusion Criteria:

* All women aged 18 and over who will receive a first allogeneic HSCT (bone marrow, peripheral blood stem cells from a related, unrelated (including cord blood) or haploidentical donor) at the CIUSSS-EMTL. Recruitment will begin when the project receives ethical approval. Recruitment period will be of 2 to 3 years.

Exclusion Criteria:

1. Those who receive a second HSCT allograft.
2. Those who receive an autologous transplant.
3. Inability to give informed consent.
4. Unable to communicate in French or English.
5. Any other reason which, according to the investigators, makes it preferable for a patient not to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All women aged 18 and over who will receive a first allogeneic HSCT
Study Population: Allotransplanted women who receive a first allogeneic stem cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Define the incidence and describe clinical presentation of vulvovaginal cGVHD after allogeneic stem cell transplants reflecting modern transplant practice. | From -1 month of transplant until +24 months after.
  Prospective history, physical exam with focus on cGVHD.

SECONDARY OUTCOMES:
Evaluate genital cGVHD treatment response | From diagnosis until 24 months post transplant
  Medical evaluation of vulvovaginal cGVHD according to NIH 2014 criteria
Evaluate the frequency of premature ovarian failure | 3, 6 and 12 months post transplant
  Percentage of patients with premature ovarian failure
Measure the incidence and prevalence of HPV infection | 3, 6 and 12 months post transplant
  Number of patients with HPV infection
Evaluate the quality of life (QoL) of allografted women | At screening and 3, 6, 12, 18 and 24 months post transplant
  Measure of QoL using FACT-BMT standardized questionnaire
Evaluate intimacy within relationships of allografted women | At screening and 6,12,18 and 24 months post transplant
  Measure of sexual health using the Personal Assessment of Intimacy within Relationships (PAIR) standardized questionnaire
Evaluate sexual function of allografted women | At screening and 6,12,18 and 24 months post transplant
  Measure of sexual health using the Female Sexual Function Index (FSFI) standardized questionnaire
Evaluate sexual distress of allografted women | At screening and 6,12,18 and 24 months post transplant
  Measure of sexual health using the Female Sexual Distress Scale-Revised (FSD-R) standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean Roy, MD, Principal Investigator — CIUSSS de l'Est de l'île de Montréal/Université de Montréal; Marie-Hélène Mayrand, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)

IPD SHARING:
Plan to Share IPD: No